CLINICAL TRIAL: NCT04664166
Title: Outcomes of Alpena Otago Telehealth Program
Brief Title: Alpena Otago Telehealth Program
Acronym: Alpena
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: Alpena Senior Citizens Center (Unknown)
Responsible Party: Principal Investigator, Min-Hui Huang, Associate professor, University of Michigan
Other Study IDs: 00184786
Record Dates: First submitted 2020-12-04; First posted 2020-12-11 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2022-01

CONDITIONS: Geriatrics; Exercise; Telemedicine
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Alpena Otago Telehealth Program — A physical therapist will use video visits to evaluate the participants and provide exercise instructions from Week 1 to Week 4. Each participant will use the Blue Marble Health in Motion app from a mobile tablet to complete the exercise guided by an avatar at their own pace after receiving the exercise instructions from the physical therapist. Participants are encouraged to exercise three days a week and 30 minutes each day using the app for 6 months. The exercise protocol based on the evidence-based Otago program includes warm up, strengthening, and balance exercise.
  3.5. Research Study Design and Data Analyses:
  Other Names: Alpena Empowered Movement Program

SUMMARY:
This project is to analyze the outcomes of the Alpena Otago Telehealth Program. The Alpena Senior Citizens Center is implementing the Otago program, an evidence-based, 6-month, home exercise program using live video chats in combination with an online exercise app, Blue Marble. We will recruit seniors who are participants of the Alpena Otago Telehealth Program to allow the study team to analyze their outcomes. The goal of the study is to examine the feasibility and efficacy of a 6-month, home-based, Otago Telehealth program for seniors in Alpena.

ELIGIBILITY:
Inclusion Criteria:

* participating in Alpena Otago telehealth program
* age >= 60 years
* ability to use a tablet
* ability to walk at home with or without a cane or walker
* ability to exercise like moving arms or legs while standing
* ability to communicate in English and follow instructions
* ability to provide the consent

Exclusion Criteria:

* advanced neurologic condition
* severe visual impairments
* falls due to syncope or dizziness

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The participants are residents living in the Alpena county and are representative of the demographics in a rural community in Michigan.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-12-04 (Actual); Study Completion 2021-12-04 (Actual)

PRIMARY OUTCOMES:
Retention rate | 6 months
  Number of participants completing the program
Fall Risk Questionnaire (FRQ) | 6 months
  The Fall Risk Questionnaire (FRQ) is a self-reported questionnaire with 12 questions for fall risk factors. Each question is rated 0 for NO (negative) and 1 for YES (positive) for fall risk factor. The sum of scores from all questions is the test score. A FRQ score >=4 indicates increased fall risk. Higher scores correspond to higher fall risk.
Activities-specific Balance Scale (ABC) | 6 months
  The Activities-specific Balance Scale (ABC) is a self-reported questionnaire of balance confidence during daily activities with 16 items. Each item is rated from 0% (NO confidence) to 100% (Completely confident) on maintaining balance for a daily task. The average of scores from all items is the test score. An ABC score <=67% indicates increased fall risk. Lower scores correspond to high worse balance confidence and higher fall risk.
PROMIS Global Health Scale v1.2 (PROMIS) | 6 months
  The PROMIS Global Health Scale v1.2 (PROMIS) is a self-reported questionnaire for health-related quality of life in physical and mental health domains.
Exercise adherence | 6 months
  Number of exercise trials completed by each participant

SECONDARY OUTCOMES:
30-Second Chair Stand Test (30CST) | 6 months
  The 30-Second Chair Stand Test (30CST) measures functional lower extremity strength.
Timed Up and Go (TUG) | 6 months
  The Timed Up and Go (TUG) measures the time it takes a person to rise up form a chair, walk 10 feet at a normal pace, turn around and sit back down in the chair with or without a mobility device. The test measures mobility.
Canadian Occupational Performance Measure (COPM) | 6 months
  The Canadian Occupational Performance Measure (COPM) is a questionnaire of difficulty in activities of daily living. Participants are asked to identify daily activities, work, or leisure activities which they want to do, need to do, or are expected to do on a typical day.
Program acceptance | 6 months
  Program acceptance is a semi-structured questionnaire about the participant's satisfaction and acceptance of program. The participants rate their opinions about the expectation, easy of use, perceived benefits and effectiveness of the exercise program on a scale of 1 to 4 (1 = "Strongly disagree", 2 = "Disagree", 3 = "Agree", 4= "Strongly Agree"). There are two open-questions about the frequency of exercise per week and suggestions for program improvement.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan-Flint, Flint, Michigan, United States

IPD SHARING:
Plan to Share IPD: No